CLINICAL TRIAL: NCT05034497
Title: A Multicenter Phase 1 Clinical Study to Determine the Maximum Tolerated Dose/Maximum Feasible Dose, Safety,& Efficacy of Single Dose Rhenium-186 NanoLiposome (186RNL) Administered Via Intraventricular Catheter for Leptomeningeal Metastases
Brief Title: Intraventricular Administration of Rhenium-186 NanoLiposome for Leptomeningeal Metastases
Acronym: ReSPECT-LM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Plus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-LM-001
Record Dates: First submitted 2021-08-23; First posted 2021-09-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Each participant will receive a single 5cc administration of 186RNL.
  At each dose level, a minimum of three to a maximum of six participants will be enrolled.
  If no dose limiting toxicity is observed in the initial three participants, then the next higher dose level cohort will open for enrollment.
  The dose escalation scheme will follow a modified Fibonacci dose escalation scheme.
  Interventions: Drug: 186RNL

INTERVENTIONS:
Drug: 186RNL — All participants will be required to have an Ommaya Reservoir and a CSF Flow Study.
  Participants will receive a single 5cc dose of 186RNL via Ommaya Reservoir.
  Other Names: Rhenium-186 NanoLiposome

SUMMARY:
This is an open-label Phase I clinical study that will administer a single dose of 186RNL via intraventricular catheter for treatment of Leptomeningeal Metastases (LM).

DETAILED DESCRIPTION:
This Phase I clinical study evaluates a single dose of 186RNL (radionuclide clinical study drug) administered through an intraventricular catheter (Ommaya reservoir) in participants with Leptomeningeal Metastases (LM).

The clinical study treatment consists of a single administered 5cc dose of 186RNL per participant.

The clinical study will include the evaluation at separate dose levels. Three to six participants may be treated at each dose.

The maximum number of participants to be enrolled in the study is 27.

The clinical study treatment will be administered, following a CSF flow study, on an outpatient basis by the clinical study physician.

Participants will be followed for up to 12 months after the clinical study drug is administered.

The U.S. Food and Drug Administration (FDA) has not approved 186RNL for this specific disease.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at time of screening.
2. Ability to understand the purposes and risks of the study and has signed a written informed consent document approved by the site-specific IRB.
3. Subject has proven and documented LM that meets the requirements for the study:

   a. Current EANO-ESMO Clinical Practice Guidelines Type 1 and 2 LM of any primary type. 2D is excluded.
4. Karnofsky performance status of 60 to 100.
5. Acceptable liver function:

   * Bilirubin 1.5 times upper limit of normal
   * AST (SGOT) and ALT (SGPT) ≤ 3.0 times upper limit of normal for subjects with normal liver
   * AST (SGOT) and ALT (SGPT) ≤ 5.0 times upper limit of normal for subjects with liver metastasis
   * Acceptable renal function with serum creatinine ≤ 2 times upper limit of normal
6. Acceptable hematologic status (without hematologic support):

   * ANC ≥ 1000 cells µL
   * Platelet count ≥ 75,000/µL
   * Hemoglobin ≥ 9.0 g/dL
7. All women of childbearing potential must have a negative serum pregnancy test at screening. Male and female subjects must agree to use effective means of contraception (for example, surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.
8. Subjects with a creatinine clearance greater than or equal to 60 mL/min (using the Cockcroft-Gault Equation) for males and females.

Exclusion Criteria:

1. The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0) Grade ≤ 1 from AEs due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study. Prior AEs due to alopecia, anemia, and lymphopenia are not required to be recovered to Grade ≤ 1 prior to 186RNL treatment, assuming other inclusion criteria are satisfied.
2. Obstructive or symptomatic communicating hydrocephalus.
3. Ventriculo-peritoneal or ventriculo-atrial shunts without programable valves or contraindications to placement of Ommaya reservoir.
4. Females of childbearing potential who are pregnant, breast feeding, or may possibly be pregnant without a negative serum pregnancy test (see inclusion criteria).
5. Serious intercurrent illness, such as progressive systemic (extra leptomeningeal) disease, clinically significant cardiac arrhythmias, uncontrolled systemic infection, symptomatic congestive heart failure or unstable angina pectoris within 3 months prior study drug, myocardial infarction, stroke, transient ischemic attack within 6 months, seizure disorder with any seizure occurring within 14 days prior to consenting or encephalopathy.
6. Active severe non hematologic organ toxicity such as renal, cardiac, hepatic, pulmonary, or gastrointestinal systemic toxicity grade 3 or above.
7. Significant coagulation abnormalities such as inherited bleeding diathesis or acquired coagulopathy with unacceptable risks of bleeding.
8. Patients who had any dose to the spinal cord or whole brain radiation therapy, regardless of when the radiation treatment was delivered. Prior, non-CNS radiation for primary tumor is allowed.
9. Systemic chemotherapeutic agents with CNS penetration (such as temozolomide, carmustine, lomustine, capecitabine, carboplatin, vinorelbine, bevacizumab, irinotecan or topotecan) are excluded if given within 14 days or 5 half-lives, whichever is shorter, prior to 186RNL treatment.

   1. If the washout period is satisfied, the patient may be enrolled, providing all other I/E criteria are satisfied.
   2. If the patient is undergoing systemic chemotherapy with CNS penetration (such as temozolomide, carmustine, lomustine, capecitabine, carboplatin, vinorelbine, bevacizumab, irinotecan or topotecan) and they develop or have progressive/persistent LM while on the agent, they may be included in the trial at the PI's discretion.
10. Systemic therapy (including investigational agents and small-molecule kinase inhibitors) is excluded if given within 14 days or 5 half-lives, whichever is shorter, prior to 186RNL treatment.

    a. If the washout period is satisfied, the patient may be enrolled, providing all other I/E criteria are satisfied.
11. Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, are excluded if given within the above timepoints prior to 186RNL treatment.

    a. If the washout period is satisfied, the patient may be enrolled, providing all other I/E criteria are satisfied.
12. Impaired CSF Flow Study, within 4 +/- 3 days of 186RNL treatment, based on study imaging and as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | 12 months
  Safety will be evaluated by the incidence of AEs and SAEs graded according CTCAE version 5.0.
Incidence of dose-limiting toxicities (DLT) | 12 months
  Maximum Tolerated Dose (MTD) will be evaluated by testing increasing doses with 3 to 6 participants in each cohort. MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants.

SECONDARY OUTCOMES:
Determination of the overall response rate (ORR) | 12 months
  Determine the overall response rate (ORR) defined as the proportion of all evaluable participants achieving a response as the best overall response at the time of progression.
Determination of the duration of response (DoR) | 12 months
  Determine the duration of response (DoR) defined as the time from first response to LM progression.
Determination of progression free survival (PFS) | 12 months
  Determine progression free survival (PFS) defined as the time from first treatment to date of LM progression or death from any cause.
Overall survival (OS) | 12 Months
  Determine the overall survival (OS) define as the time from first treatment to date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, PhD, Principal Investigator — The Cancer Therapy and Research Center at UTSHSCSA
Locations (6):
- United States (6):
  - Northwestern Memorial Hospital Olson Pavilion, Chicago, Illinois
  - Northshore University Hospital, Manhasset, New York
  - Lenox Hill Hospital, New York, New York
  - Ohio State University Hospital, Columbus, Ohio
  - Universiy of Texas Southwestern Medical Center, Dallas, Texas
  - UT Health Science Center San Antonio / Mays Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No